CLINICAL TRIAL: NCT01196975
Title: Immunogenicity, Reactogenicity and Safety of GSK Biologicals' Quadrivalent Influenza Vaccine FLU Q-QIV (GSK2282512A) When Administered Intramuscularly to Adults 18 Years of Age and Older
Brief Title: A Study to Evaluate the Safety and Immunogenicity of GSK Biologicals' Seasonal Influenza Vaccine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 112963
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Results first posted 2012-12-24 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2016-09

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- GSK2282512A 1 Group (Experimental): Subjects received at Day 0 one dose of the GSK2282512A vaccine, Lot 1. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Quadrivalent seasonal influenza vaccine GSK2282512A
- GSK2282512A 2 Group (Experimental): Subjects received at Day 0 one dose of the GSK2282512A vaccine, Lot 2. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Quadrivalent seasonal influenza vaccine GSK2282512A
- GSK2282512A 3 Group (Experimental): Subjects received at Day 0 one dose of the GSK2282512A vaccine, Lot 3. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Quadrivalent seasonal influenza vaccine GSK2282512A
- Victoria Strain FluLaval Group (Active Comparator): Subjects received at Day 0 one dose of FluLaval®-VB vaccine containing the Victoria B flu strain. The FluLaval®-VB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: FluLavalTM-VB
- Yamagata Strain FluLaval Group (Active Comparator): Subjects received at Day 0 one dose of FluLaval®-YB vaccine containing the Yamagata B flu strain. The FluLaval®-YB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: FluLavalTM-YB

INTERVENTIONS:
Biological: Quadrivalent seasonal influenza vaccine GSK2282512A — Single intramuscular dose
  Other Names: GSK2282512A
  Arms: GSK2282512A 1 Group; GSK2282512A 2 Group; GSK2282512A 3 Group
Biological: FluLavalTM-VB — Single intramuscular dose
  Other Names: FluLavalTM containing the Victoria B flu strain; FluLaval®-VB; Victoria Strain FluLaval vaccine
  Arms: Victoria Strain FluLaval Group
Biological: FluLavalTM-YB — Single intramuscular dose
  Other Names: FluLavalTM containing the Yamagata B flu strain; FluLaval®-YB
  Arms: Yamagata Strain FluLaval Group

SUMMARY:
This study is designed to test the immunogenicity and safety of an investigational influenza vaccine, in adults compared to two other influenza vaccines.

This study will also evaluate the lot-to-lot consistency of three vaccine lots.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol
* A male or female 18 years of age or older, in stable health, as established by medical history and physical examination before entering into the study.
* Written informed consent obtained from the subject.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line, or mobile, but NOT a pay phone or other multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* - has practiced adequate contraception for 30 days prior to vaccination, and
* - has a negative pregnancy test on the day of vaccination, and
* - has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of an investigational / non-registered product other than the study vaccines within 30 days before study vaccination or planned use during study period.
* Planned administration or administration of a licensed vaccine within 30 days before study vaccination.
* Prior receipt of 2010/2011 influenza vaccine.
* Receipt of any investigational or approved influenza vaccine within six months of the first study visit.
* Any known or suspected allergy to any constituent of influenza vaccines ; a history of anaphylactic-type reaction to constituent of vaccine; or a history of severe adverse reaction to a previous influenza vaccine.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* History of Guillain-Barre syndrome within 6 weeks of receipt of prior inactivated influenza virus vaccine.
* Presence or evidence of substance abuse or of neurological or psychiatric diagnoses which, even if clinically stable, are deemed by the investigator to render the potential subject unable / unlikely to provide accurate safety reports.
* Acute, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, based on history and physical examination.
* Presence of significant uncontrolled chronic medical or neuropsychiatric illness, based on history and physical examination
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Any significant disorder of coagulation or treatment with Coumadin derivatives or heparin
* Chronic administration of immunosuppressants or other immune-modifying drugs within 3 months prior to the first vaccine/product dose.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Fever at the time of enrolment.
* Acute disease at the time of enrolment
* Any other condition which, in the opinion of the Investigator, prevents the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1707 (Actual)
Dates: Start 2010-10-01; Primary Completion 2011-01-25 (Actual); Study Completion 2011-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (6):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Jefferson Hills, Pennsylvania
  - GSK Investigational Site, Wenatchee, Washington
- Canada (3):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Québec, Quebec
- Mexico (3):
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Estado de México

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Tinoco JC, Pavia-Ruz N, Cruz-Valdez A, Aranza Doniz C, Chandrasekaran V, Dewe W, Liu A, Innis BL, Jain VK. Immunogenicity, reactogenicity, and safety of inactivated quadrivalent influenza vaccine candidate versus inactivated trivalent influenza vaccine in healthy adults aged >/=18 years: a phase III, randomized trial. Vaccine. 2014 Mar 14;32(13):1480-7. doi: 10.1016/j.vaccine.2014.01.022. Epub 2014 Jan 28. PMID 24486352
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 112963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112963 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1703 of the 1707 subjects enrolled in the study were actually administered vaccination. The other 4 subjects were not vaccinated due to failing at meeting protocol specific criteria.
Pre-assignment Details: For some outcome measures, the subjects receiving the GSK2282512A vaccine, from Lot 1, 2 or 3, were pooled into one larger pooled group, the GSK2282512A Group, and/or groups were stratified into the 4 age categories: 18 to 60 years (18-60Y), 61 years and older (≥61Y), 18 to 64 years (18-64Y), and 65 years and older (≥ 65Y).
Period: Overall Study
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Started | 423 | 424 | 425 | 213 | 218
Completed | 408 | 415 | 420 | 207 | 205
Not Completed | 15 | 9 | 5 | 6 | 13
Not completed — Adverse Event | 2 | 2 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 11 | 6 | 5 | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group | Total
Number analyzed (Participants) | 423 | 424 | 425 | 213 | 218 | 1703
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (19.49) | 50.4 (19.07) | 49.8 (20.10) | 50.8 (18.58) | 49.6 (19.34) | 50.1 (19.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 264 | 266 | 125 | 138 | 1044
  Male | 172 | 160 | 159 | 88 | 80 | 659

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was 1:10. Antibodies assessed were antibodies against the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 (FLO) flu strains. Results for Day 21 for the subjects in the GSK2282512A Group are the results specific to this primary outcome measure.
Time Frame: At Day 0 (D0) and at Day 21 (D21) post vaccination.
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all vaccinated and eligible subjects for whom data concerning Immunogenicity outcomes variables were available and for whom assay results were available for antibodies against at least one study vaccine component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- GSK2282512A Group: Subjects received at Day 0 one dose of the GSK2282512A vaccine, from Lot 1, 2 or 3. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Yamagata Strain FluLaval Group: Yamagata Strain FluLaval Group - Subjects received at Day 0 one dose of FluLaval®-YB vaccine containing the Yamagata B flu strain. The FluLaval®-YB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | GSK2282512A Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 1246 | 204 | 211
Titer
  H1N1, D0: number analyzed (Participants) | 1238 | 204 | 211
  H1N1, D0 | 16.9 [15.7 to 18.2] | 19.1 [15.8 to 23.1] | 16.5 [13.9 to 19.6]
  H1N1, D21: number analyzed (Participants) | 1246 | 204 | 210
  H1N1, D21 | 204.6 [190.4 to 219.9] | 176.0 [149.1 to 207.7] | 149.0 [122.9 to 180.7]
  H3N1, D0: number analyzed (Participants) | 1238 | 204 | 211
  H3N1, D0 | 16.0 [15.0 to 17.1] | 13.9 [11.8 to 16.4] | 14.9 [12.7 to 17.5]
  H3N1, D21: number analyzed (Participants) | 1245 | 204 | 211
  H3N1, D21 | 125.4 [117.4 to 133.9] | 147.5 [124.1 to 175.2] | 141.0 [118.1 to 168.3]
  BRI, D0: number analyzed (Participants) | 1240 | 203 | 211
  BRI, D0 | 27.9 [26.0 to 30.0] | 29.4 [24.7 to 35.0] | 26.7 [22.8 to 31.4]
  BRI, D21: number analyzed (Participants) | 1246 | 204 | 210
  BRI, D21 | 177.7 [167.8 to 188.1] | 135.9 [118.1 to 156.5] | 71.9 [61.3 to 84.2]
  FLO, D0: number analyzed (Participants) | 1241 | 204 | 211
  FLO, D0 | 76.2 [71.1 to 81.5] | 68.1 [58.5 to 79.2] | 70.3 [59.8 to 82.6]
  FLO, D21 | 399.7 [378.1 to 422.6] | 176.9 [153.8 to 203.5] | 306.6 [266.2 to 353.3]

2. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease by Age Strata
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was 1:10. Antibodies assessed were antibodies against the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 flu strains. Subjects were assessed according to 2 age categories, 18-64Y and ≥ 65Y.
Time Frame: At Day 0 (D0) and at Day 21 (D21) post vaccination.
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all vaccinated and eligible subjects for whom data concerning Immunogenicity outcomes variables were available and for whom assay results were available for antibodies against at least one study vaccine component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- GSK2282512A 18-64Y Group: Subjects aged between 18 and up to 64 years inclusive at the time of vaccination received at Day 0 one dose of the GSK2282512A vaccine, from Lot 1, 2 or 3. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- GSK2282512A ≥ 65Y Group: Subjects aged 65 years or above at the time of vaccination received at Day 0 one dose of the GSK2282512A vaccine, from Lot 1, 2 or 3. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Victoria Strain FluLaval 18-64Y Group: Subjects aged between 18 and up to 64 years inclusive at the time of vaccination received at Day 0 one dose of FluLaval®-VB vaccine containing the Victoria B flu strain. The FluLaval®-VB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Victoria Strain FluLaval ≥ 65Y Group: Subjects aged 65 years or above at the time of vaccination received at Day 0 one dose of FluLaval®-VB vaccine containing the Victoria B flu strain. The FluLaval®-VB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Yamagata Strain FluLaval 18-64Y Group: Subjects aged between 18 and up to 64 years inclusive at the time of vaccination received at Day 0 one dose of FluLaval®-YB vaccine containing the Yamagata B flu strain. The FluLaval®-YB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Yamagata Strain FluLaval ≥ 65Y Group: Subjects aged 65 years or above at the time of vaccination received at Day 0 one dose of FluLaval®-YB vaccine containing the Yamagata B flu strain. The FluLaval®-YB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | GSK2282512A 18-64Y Group | GSK2282512A ≥ 65Y Group | Victoria Strain FluLaval 18-64Y Group | Victoria Strain FluLaval ≥ 65Y Group | Yamagata Strain FluLaval 18-64Y Group | Yamagata Strain FluLaval ≥ 65Y Group
Number analyzed (Participants) | 849 | 397 | 136 | 68 | 144 | 68
titer
  H1N1, D0: number analyzed (Participants) | 844 | 394 | 136 | 68 | 144 | 67
  H1N1, D0 | 19.0 [17.4 to 20.9] | 13.2 [11.7 to 14.7] | 20.3 [16.0 to 25.8] | 16.8 [12.3 to 22.9] | 18.7 [15.0 to 23.2] | 12.6 [9.6 to 16.5]
  H1N1, D21: number analyzed (Participants) | 849 | 397 | 136 | 68 | 143 | 67
  H1N1, D21 | 289.4 [267.9 to 312.7] | 97.4 [85.9 to 110.5] | 236.9 [199.7 to 281.1] | 97.1 [70.3 to 134.1] | 198.5 [161.7 to 243.7] | 80.8 [55.1 to 118.5]
  H3N1, D0: number analyzed (Participants) | 844 | 394 | 136 | 68 | 144 | 67
  H3N1, D0 | 15.2 [14.0 to 16.6] | 17.8 [15.9 to 19.9] | 15.0 [12.1 to 18.4] | 12.0 [9.1 to 15.8] | 14.8 [12.1 to 18.1] | 15.1 [11.6 to 19.7]
  H3N1, D21: number analyzed (Participants) | 849 | 396 | 136 | 68 | 144 | 67
  H3N1, D21 | 136.1 [125.9 to 147.2] | 105.1 [93.4 to 118.3] | 176.3 [144.3 to 215.4] | 103.2 [75.1 to 141.8] | 173.6 [142.5 to 211.6] | 90.1 [63.8 to 127.3]
  BRI, D0: number analyzed (Participants) | 843 | 397 | 135 | 68 | 144 | 67
  BRI, D0 | 21.7 [19.9 to 23.7] | 47.9 [42.8 to 53.5] | 23.8 [19.1 to 29.6] | 44.7 [34.1 to 58.6] | 22.8 [18.7 to 27.8] | 37.6 [28.8 to 49.1]
  BRI, D21: number analyzed (Participants) | 849 | 397 | 136 | 68 | 143 | 67
  BRI, D21 | 199.3 [185.9 to 213.6] | 139.0 [126.2 to 153.1] | 157.2 [131.5 to 187.9] | 101.6 [81.8 to 126.1] | 75.1 [61.2 to 92.2] | 65.4 [51.3 to 83.4]
  FLO, D0: number analyzed (Participants) | 844 | 397 | 136 | 68 | 144 | 67
  FLO, D0 | 70.7 [64.8 to 77.2] | 89.1 [80.2 to 98.9] | 66.1 [54.3 to 80.4] | 72.2 [57.2 to 91.2] | 67.6 [54.8 to 83.4] | 76.3 [59.9 to 97.3]
  FLO, D21: number analyzed (Participants) | 849 | 397 | 136 | 68 | 144 | 67
  FLO, D21 | 475.3 [444.2 to 508.5] | 276.1 [252.8 to 301.5] | 204.9 [171.3 to 245.0] | 131.8 [107.1 to 162.3] | 406.1 [347.3 to 474.9] | 167.7 [132.0 to 212.9]

3. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease by Age Strata
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was 1:10. Antibodies assessed were antibodies against the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 flu strains. Subjects were assessed according to 2 age categories, 18-60Y and ≥ 61Y.
Time Frame: At Day 0 (D0), and at Day 21 (D21) and Day 180 (D180) post vaccination.
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for persistence, which included all vaccinated subjects who had not received a vaccine forbidden in the protocol with available assay results for assessed antibodies in Day 180 blood samples.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- GSK2282512A 18-60Y Group: Subjects aged between 18 and up to 60 years inclusive at the time of vaccination received at Day 0 one dose of the GSK2282512A vaccine, from Lot 1, 2 or 3. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- GSK2282512A ≥ 61Y Group: Subjects aged 61 years or above at the time of vaccination received at Day 0 one dose of the GSK2282512A vaccine, from Lot 1, 2 or 3. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Victoria Strain FluLaval 18-60Y Group: Subjects aged between 18 and up to 60 years inclusive at the time of vaccination received at Day 0 one dose of FluLaval®-VB vaccine containing the Victoria B flu strain. The FluLaval®-VB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Victoria Strain FluLaval ≥ 61Y Group: Subjects aged 61 years or above at the time of vaccination received at Day 0 one dose of FluLaval®-VB vaccine containing the Victoria B flu strain. The FluLaval®-VB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Yamagata Strain FluLaval 18-60Y Group: Subjects aged between 18 and up to 60 years inclusive at the time of vaccination received at Day 0 one dose of FluLaval®-YB vaccine containing the Yamagata B flu strain. The FluLaval®-YB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
- Yamagata Strain FluLaval ≥ 61Y Group: Subjects aged 61 years or above at the time of vaccination received at Day 0 one dose of FluLaval®-YB vaccine containing the Yamagata B flu strain. The FluLaval®-YB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | GSK2282512A 18-60Y Group | GSK2282512A ≥ 61Y Group | Victoria Strain FluLaval 18-60Y Group | Victoria Strain FluLaval ≥ 61Y Group | Yamagata Strain FluLaval 18-60Y Group | Yamagata Strain FluLaval ≥ 61Y Group
Number analyzed (Participants) | 122 | 135 | 17 | 20 | 22 | 20
titer
  H1N1, D0 | 23.1 [17.9 to 29.8] | 12.0 [9.9 to 14.5] | 22.6 [11.6 to 44.0] | 18.7 [8.7 to 39.9] | 17.9 [10.0 to 32.1] | 10.2 [6.1 to 17.0]
  H1N1, D21 | 302.4 [245.8 to 372.0] | 105.0 [83.6 to 131.9] | 369.1 [216.2 to 630.0] | 132.2 [64.5 to 270.7] | 187.4 [110.4 to 318.2] | 81.4 [34.2 to 194.1]
  H1N1, D180 | 97.9 [80.3 to 119.3] | 29.1 [23.4 to 36.2] | 104.2 [57.0 to 190.5] | 55.6 [29.3 to 105.6] | 57.5 [33.2 to 99.4] | 34.8 [16.2 to 74.8]
  H3N1, D0 | 15.5 [12.3 to 19.4] | 17.9 [14.7 to 21.8] | 12.0 [7.3 to 19.7] | 16.8 [9.1 to 30.9] | 12.7 [7.7 to 20.7] | 17.1 [9.9 to 29.6]
  H3N1, D21: number analyzed (Participants) | 122 | 134 | 17 | 20 | 22 | 20
  H3N1, D21 | 123.2 [100.4 to 151.2] | 119.8 [97.6 to 147.0] | 163.3 [103.0 to 258.8] | 168.4 [82.1 to 345.6] | 175.9 [110.7 to 279.3] | 157.2 [92.3 to 267.9]
  H3N1, D180 | 40.9 [33.5 to 49.9] | 43.3 [36.7 to 51.1] | 46.1 [31.8 to 67.0] | 46.7 [27.6 to 79.0] | 63.0 [39.5 to 100.8] | 60.6 [35.1 to 104.6]
  BRI, D0 | 22.9 [18.3 to 28.6] | 41.1 [33.9 to 49.8] | 30.7 [16.1 to 58.6] | 42.9 [25.4 to 72.3] | 17.9 [11.7 to 27.3] | 32.5 [18.0 to 58.6]
  BRI, D21 | 193.0 [161.0 to 231.4] | 167.2 [141.6 to 197.3] | 180.9 [120.9 to 270.7] | 109.3 [77.7 to 153.6] | 53.9 [31.0 to 93.6] | 74.7 [44.7 to 124.9]
  BRI, D180 | 112.8 [94.1 to 135.3] | 127.0 [109.1 to 147.8] | 130.5 [91.8 to 185.4] | 102.0 [78.8 to 132.0] | 59.3 [36.9 to 95.4] | 79.9 [49.8 to 128.5]
  FLO, D0 | 75.4 [59.3 to 95.8] | 79.2 [65.5 to 95.7] | 92.3 [54.5 to 156.4] | 93.5 [54.0 to 161.7] | 60.3 [38.7 to 93.9] | 78.6 [41.6 to 148.3]
  FLO, D21 | 485.8 [407.3 to 579.5] | 334.3 [288.9 to 386.8] | 204.4 [134.8 to 310.0] | 187.0 [138.5 to 252.3] | 405.3 [273.8 to 600.0] | 180.6 [101.4 to 321.7]
  FLO, D180 | 311.9 [261.7 to 371.7] | 209.5 [183.0 to 239.8] | 177.3 [120.5 to 260.9] | 160.1 [108.8 to 235.6] | 320.1 [207.8 to 492.9] | 174.3 [104.3 to 291.2]

4. Secondary Outcome: Number of Subjects With Medically-attended Adverse Events (MAEs)
Description: Medically-attended adverse events (MAEs) were non-serious and serious events leading to an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits. If a medically-attended adverse event was leading to hospitalization (or met any other serious adverse event [SAE] criterion), it was reported as SAE.
Time Frame: From the beginning of the study until study end (from Day 0 to Day 180)
Population: The analysis was performed on the Total Vaccinated cohort, on subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 423 | 424 | 425 | 213 | 218
Participants | 129 | 101 | 100 | 51 | 64

5. Secondary Outcome: Number of Subjects With Related Medically-attended Adverse Events (MAEs)
Description: Medically-attended adverse events (MAEs) were non-serious and serious events leading to an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits. If a medically-attended adverse event was leading to hospitalization (or met any other serious adverse event [SAE] criterion), it was reported as SAE. Related MAE = MAE assessed by the investigator to be causally related to vaccination. Relationship to vaccination was not computed for MAEs.
Time Frame: From the beginning of the study until study end (from Day 0 to Day 180) .
Population: The analysis was performed on the Total Vaccinated cohort, on subjects with available results.
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Subjects With Any and Related Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of adverse events that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. Related pIMD = pIMD assessed by the investigator to be causally related to vaccination.
Time Frame: From the beginning of the study until study end (from Day 0 to Day 180) .
Population: The analysis was performed on the Total Vaccinated cohort, on subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 423 | 424 | 425 | 213 | 218
Participants
  Subject(s) with Any pIMD(s) | 1 | 1 | 1 | 0 | 1
  Subject(s) with Related pIMD(s) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From the beginning of the study until study end (from Day 0 to Day 180)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 423 | 424 | 425 | 213 | 218
Participants
  Subject(s) with Any SAE(s) | 15 | 13 | 7 | 3 | 7
  Subject(s) with Related SAE(s) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease by Age Strata
Description: as for outcome 2
Time Frame: At Day 0 (D0), and at Day 21 (D21) and Day 180 (D180) post vaccination.
Population: The analysis was performed on the According-To-Protocol cohort for persistence, which included all vaccinated subjects who had not received a vaccine forbidden in the protocol, and with available assay results at Day 180 for assessed antibodies.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK2282512A 18-64Y Group | GSK2282512A ≥ 65Y Group | Victoria Strain FluLaval 18-64Y Group | Victoria Strain FluLaval ≥ 65Y Group | Yamagata Strain FluLaval 18-64Y Group | Yamagata Strain FluLaval ≥ 65Y Group
Number analyzed (Participants) | 131 | 126 | 18 | 19 | 23 | 19
Titer
  H1N1, D0 | 22.7 [17.8 to 29.0] | 11.6 [9.6 to 14.2] | 23.3 [12.4 to 43.7] | 17.9 [8.1 to 39.8] | 18.0 [10.3 to 31.4] | 9.8 [5.7 to 16.8]
  H1N1, D21 | 293.3 [240.7 to 357.3] | 100.5 [79.1 to 127.7] | 339.0 [199.0 to 577.6] | 135.7 [63.7 to 289.2] | 180.6 [108.4 to 300.8] | 81.5 [32.5 to 204.3]
  H1N1, D180 | 95.5 [79.1 to 115.3] | 27.4 [21.8 to 34.4] | 98.8 [55.5 to 176.0] | 56.6 [28.7 to 111.4] | 56.6 [33.5 to 95.4] | 34.5 [15.4 to 77.6]
  H3N1, D0 | 15.3 [12.2 to 19.1] | 18.4 [15.1 to 22.3] | 13.3 [8.0 to 22.4] | 15.5 [8.3 to 28.8] | 12.2 [7.5 to 19.6] | 18.2 [10.4 to 32.2]
  H3N1, D21: number analyzed (Participants) | 131 | 125 | 18 | 19 | 23 | 19
  H3N1, D21 | 115.0 [93.2 to 141.9] | 128.6 [105.4 to 156.8] | 163.1 [105.8 to 251.3] | 168.9 [79.0 to 361.3] | 175.1 [112.7 to 272.2] | 157.1 [89.4 to 276.0]
  H3N1, D180 | 41.3 [34.0 to 50.0] | 43.1 [36.3 to 51.0] | 49.4 [33.8 to 72.2] | 43.8 [25.6 to 74.9] | 61.9 [39.5 to 96.9] | 61.9 [34.8 to 110.1]
  BRI, D0 | 23.1 [18.6 to 28.6] | 42.5 [34.8 to 51.8] | 29.9 [16.3 to 55.1] | 44.6 [25.9 to 77.0] | 19.7 [12.6 to 30.8] | 29.9 [16.5 to 54.2]
  BRI, D21 | 183.6 [154.3 to 218.6] | 174.3 [146.6 to 207.1] | 166.4 [109.6 to 252.5] | 115.2 [81.9 to 162.0] | 56.5 [33.1 to 96.5] | 71.8 [41.9 to 122.8]
  BRI, D180 | 111.1 [93.6 to 131.8] | 130.2 [111.0 to 152.7] | 124.6 [88.4 to 175.7] | 105.2 [80.8 to 137.0] | 63.8 [39.6 to 102.9] | 74.3 [46.2 to 119.5]
  FLO, D0 | 78.5 [62.4 to 98.8] | 76.1 [62.6 to 92.6] | 98.9 [59.1 to 165.6] | 87.6 [50.0 to 153.7] | 64.8 [41.4 to 101.5] | 73.0 [38.0 to 140.0]
  FLO, D21 | 473.4 [399.7 to 560.6] | 334.4 [287.4 to 389.1] | 209.5 [141.3 to 310.8] | 181.7 [133.2 to 248.0] | 401.2 [275.9 to 583.3] | 175.3 [95.5 to 321.6]
  FLO, D180 | 314.1 [266.4 to 370.4] | 202.1 [175.6 to 232.7] | 190.4 [128.6 to 281.9] | 148.8 [102.3 to 216.6] | 329.9 [217.6 to 500.1] | 162.8 [96.6 to 274.2]

9. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition titer ≥ 1:40. The 4 assessed influenza strains were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N1), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 (FLO) flu strains
Time Frame: At Day 0 (D0) and at Day 21 (D21) after vaccination.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- GSK2282512A Group: Subjects received at Day 0 one dose of the GSK2282512A vaccine, Lot 1, 2 or 3. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | GSK2282512A Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 1246 | 204 | 211
Participants
  H1N1, D0: number analyzed (Participants) | 1238 | 204 | 211
  H1N1, D0 | 423 | 78 | 63
  H1N1, D21: number analyzed (Participants) | 1246 | 204 | 210
  H1N1, D21 | 1168 | 189 | 182
  H3N1, D0: number analyzed (Participants) | 1238 | 204 | 211
  H3N1, D0 | 385 | 55 | 64
  H3N1, D21: number analyzed (Participants) | 1245 | 204 | 211
  H3N1, D21 | 1130 | 188 | 193
  BRI, D0: number analyzed (Participants) | 1240 | 204 | 211
  BRI, D0 | 635 | 103 | 98
  BRI, D21: number analyzed (Participants) | 1246 | 204 | 210
  BRI, D21 | 1201 | 193 | 167
  FLO, D0: number analyzed (Participants) | 1241 | 204 | 211
  FLO, D0 | 997 | 162 | 168
  FLO, D21 | 1244 | 200 | 207

10. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease by Age Strata
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition titer ≥ 1:40. The 4 assessed influenza strains were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N1), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 (FLO) flu strains. Subjects were assessed according to 2 age categories, 18-60Y and ≥ 61Y.
Time Frame: At Day 0 (D0) and at Day 21 (D21) after vaccination.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 18-60Y Group | GSK2282512A ≥ 61Y Group | Victoria Strain FluLaval 18-60Y Group | Victoria Strain FluLaval ≥ 61Y Group | Yamagata Strain FluLaval 18-60Y Group | Yamagata Strain FluLaval ≥ 61Y Group
Number analyzed (Participants) | 780 | 466 | 127 | 77 | 135 | 76
Participants
  H1N1, D0: number analyzed (Participants) | 775 | 463 | 127 | 77 | 135 | 76
  H1N1, D0 | 309 | 114 | 51 | 27 | 50 | 13
  H1N1, D21: number analyzed (Participants) | 780 | 466 | 127 | 77 | 135 | 75
  H1N1, D21 | 765 | 403 | 125 | 64 | 127 | 55
  H3N1, D0: number analyzed (Participants) | 775 | 463 | 127 | 77 | 135 | 76
  H3N1, D0 | 229 | 156 | 38 | 17 | 40 | 24
  H3N1, D21: number analyzed (Participants) | 780 | 465 | 127 | 77 | 135 | 76
  H3N1, D21 | 726 | 404 | 122 | 66 | 130 | 63
  BRI, D0: number analyzed (Participants) | 774 | 466 | 126 | 77 | 135 | 76
  BRI, D0 | 338 | 297 | 52 | 51 | 53 | 45
  BRI, D21: number analyzed (Participants) | 780 | 466 | 127 | 77 | 135 | 75
  BRI, D21 | 760 | 441 | 121 | 72 | 107 | 60
  FLO, D0: number analyzed (Participants) | 775 | 466 | 127 | 77 | 135 | 76
  FLO, D0 | 591 | 406 | 99 | 63 | 105 | 63
  FLO, D21 | 779 | 465 | 125 | 75 | 134 | 73

11. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease by Age Strata
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition titer ≥ 1:40. The 4 assessed influenza strains were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N1), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 (FLO) flu strains. Subjects were assessed according to 2 age categories, 18-64Y and ≥ 65Y.
Time Frame: At Day 0 (D0) and at Day 21 (D21) after vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 18-64Y Group | GSK2282512A ≥ 65Y Group | Victoria Strain FluLaval 18-64Y Group | Victoria Strain FluLaval ≥ 65Y Group | Yamagata Strain FluLaval 18-64Y Group | Yamagata Strain FluLaval ≥ 65Y Group
Number analyzed (Participants) | 849 | 397 | 136 | 68 | 144 | 67
Participants
  H1N1, D0: number analyzed (Participants) | 844 | 394 | 136 | 68 | 144 | 67
  H1N1, D0 | 330 | 93 | 55 | 23 | 51 | 12
  H1N1, D21: number analyzed (Participants) | 849 | 397 | 136 | 68 | 143 | 67
  H1N1, D21 | 830 | 338 | 134 | 55 | 132 | 50
  H3N1, D0: number analyzed (Participants) | 844 | 394 | 136 | 68 | 144 | 67
  H3N1, D0 | 251 | 134 | 40 | 15 | 42 | 22
  H3N1, D21: number analyzed (Participants) | 849 | 396 | 136 | 68 | 144 | 67
  H3N1, D21 | 784 | 346 | 129 | 59 | 137 | 56
  BRI, D0: number analyzed (Participants) | 843 | 397 | 135 | 68 | 144 | 67
  BRI, D0 | 366 | 269 | 55 | 48 | 59 | 39
  BRI, D21: number analyzed (Participants) | 849 | 397 | 136 | 68 | 143 | 67
  BRI, D21 | 826 | 375 | 130 | 63 | 114 | 53
  FLO, D0: number analyzed (Participants) | 844 | 397 | 136 | 68 | 144 | 67
  FLO, D0 | 650 | 347 | 105 | 57 | 112 | 56
  FLO, D21 | 848 | 396 | 134 | 66 | 143 | 64

12. Secondary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza by Age Strata
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥1:40, or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 4 assessed influenza strains were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N1), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 (FLO) flu strains. Subjects were assessed according to 2 age categories, 18-64Y and ≥ 65Y.
Time Frame: At Day 21 (D21) after vaccination.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 18-64Y Group | GSK2282512A ≥ 65Y Group | Victoria Strain FluLaval 18-64Y Group | Victoria Strain FluLaval ≥ 65Y Group | Yamagata Strain FluLaval 18-64Y Group | Yamagata Strain FluLaval ≥ 65Y Group
Number analyzed (Participants) | 844 | 397 | 136 | 68 | 144 | 67
Participants
  H1N1, D21: number analyzed (Participants) | 844 | 394 | 136 | 68 | 143 | 67
  H1N1, D21 | 667 | 255 | 101 | 35 | 102 | 36
  H3N1, D21: number analyzed (Participants) | 844 | 393 | 136 | 68 | 144 | 67
  H3N1, D21 | 584 | 239 | 104 | 45 | 109 | 40
  BRI, D21: number analyzed (Participants) | 843 | 397 | 135 | 68 | 143 | 67
  BRI, D21 | 561 | 124 | 80 | 19 | 52 | 10
  FLO, D21 | 533 | 147 | 55 | 13 | 90 | 17

13. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease by Age Strata
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0 (i.e. the geometric mean of the within-subject ratios of the Day 21 reciprocal HI titer to the Day 0 reciprocal HI titer). The 4 assessed influenza strains were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N1), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 (FLO) flu strains. Subjects were assessed according to 2 age categories, 18-64Y and ≥ 65Y.
Time Frame: At Day 21 (D21) after vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK2282512A 18-64Y Group | GSK2282512A ≥ 65Y Group | Victoria Strain FluLaval 18-64Y Group | Victoria Strain FluLaval ≥ 65Y Group | Yamagata Strain FluLaval 18-64Y Group | Yamagata Strain FluLaval ≥ 65Y Group
Number analyzed (Participants) | 844 | 397 | 136 | 68 | 144 | 67
Titer
  SCF - H1N1, D21: number analyzed (Participants) | 844 | 394 | 136 | 68 | 143 | 67
  SCF - H1N1, D21 | 15.2 [13.7 to 16.9] | 7.4 [6.4 to 8.4] | 11.7 [9.0 to 15.1] | 5.8 [4.0 to 8.3] | 10.5 [8.2 to 13.4] | 6.4 [4.3 to 9.5]
  SCF - H3N1, D21: number analyzed (Participants) | 844 | 393 | 136 | 68 | 144 | 67
  SCF - H3N1, D21 | 8.9 [8.1 to 9.8] | 5.9 [5.2 to 6.7] | 11.8 [9.2 to 15.1] | 8.6 [5.9 to 12.4] | 11.7 [9.1 to 15.1] | 6.0 [4.3 to 8.3]
  SCF - BRI, D21: number analyzed (Participants) | 843 | 397 | 135 | 68 | 143 | 67
  SCF - BRI, D21 | 9.2 [8.3 to 10.1] | 2.9 [2.6 to 3.2] | 6.5 [5.1 to 8.3] | 2.3 [1.8 to 2.9] | 3.3 [2.7 to 4.1] | 1.7 [1.4 to 2.2]
  SCF - FLO, D21 | 6.7 [6.1 to 7.4] | 3.1 [2.8 to 3.4] | 3.1 [2.6 to 3.7] | 1.8 [1.5 to 2.3] | 6.0 [4.8 to 7.5] | 2.2 [1.8 to 2.7]

14. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease by Age Strata
Description: as for outcome 3
Time Frame: At Day 0 (D0) and at Day 21 (D21) post vaccination.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | GSK2282512A 18-60Y Group | GSK2282512A ≥ 61Y Group | Victoria Strain FluLaval 18-60Y Group | Victoria Strain FluLaval ≥ 61Y Group | Yamagata Strain FluLaval 18-60Y Group | Yamagata Strain FluLaval ≥ 61Y Group
Number analyzed (Participants) | 780 | 466 | 127 | 77 | 135 | 76
titer
  H1N1, D0: number analyzed (Participants) | 775 | 463 | 127 | 77 | 135 | 76
  H1N1, D0 | 19.5 [17.7 to 21.5] | 13.4 [12.0 to 14.9] | 20.7 [16.1 to 26.6] | 16.6 [12.4 to 22.3] | 19.3 [15.4 to 24.2] | 12.5 [9.7 to 16.1]
  H1N1, D21: number analyzed (Participants) | 780 | 466 | 127 | 77 | 135 | 75
  H1N1, D21 | 306.9 [283.3 to 332.5] | 103.8 [92.6 to 116.3] | 248.3 [207.8 to 296.6] | 99.7 [74.7 to 133.2] | 212.2 [175.2 to 257.0] | 78.9 [54.0 to 115.3]
  H3N1, D0: number analyzed (Participants) | 775 | 463 | 127 | 77 | 135 | 76
  H3N1, D0 | 15.4 [14.1 to 16.8] | 17.1 [15.4 to 19.0] | 15.4 [12.4 to 19.1] | 11.8 [9.1 to 15.2] | 14.8 [12.0 to 18.3] | 15.0 [11.7 to 19.2]
  H3N1, D21: number analyzed (Participants) | 780 | 465 | 127 | 77 | 135 | 76
  H3N1, D21 | 141.0 [130.1 to 152.9] | 102.9 [92.2 to 114.8] | 187.0 [152.0 to 229.9] | 99.7 [74.7 to 133.1] | 178.2 [145.9 to 217.7] | 93.0 [67.1 to 128.9]
  BRI, D0: number analyzed (Participants) | 774 | 466 | 126 | 77 | 135 | 76
  BRI, D0 | 21.6 [19.7 to 23.7] | 42.8 [38.4 to 47.7] | 23.9 [19.1 to 29.9] | 41.3 [31.6 to 53.8] | 21.6 [17.7 to 26.5] | 38.9 [30.3 to 50.0]
  BRI, D21: number analyzed (Participants) | 780 | 466 | 127 | 77 | 135 | 75
  BRI, D21 | 204.8 [190.5 to 220.2] | 140.1 [128.1 to 153.1] | 164.4 [137.0 to 197.4] | 99.3 [80.7 to 122.0] | 73.3 [59.2 to 90.7] | 69.3 [55.1 to 87.3]
  FLO, D0: number analyzed (Participants) | 775 | 466 | 127 | 77 | 135 | 76
  FLO, D0 | 70.5 [64.3 to 77.2] | 86.7 [78.6 to 95.6] | 66.4 [54.0 to 81.7] | 70.8 [57.2 to 87.7] | 64.3 [52.5 to 81.3] | 80.0 [63.7 to 100.4]
  FLO, D21 | 493.1 [459.3 to 529.3] | 281.4 [259.6 to 304.9] | 211.4 [175.0 to 255.3] | 131.9 [109.2 to 159.1] | 413.7 [351.2 to 487.2] | 180.2 [144.3 to 224.9]

15. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The reference cut-off value was 1:10. Antibodies assessed were antibodies against the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N2), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 flu strains.
Time Frame: At Day 0 (D0), and at Day 21 (D21) and Day 180 (D180) post vaccination.
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK2282512A Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 257 | 37 | 42
Titer
  H1N1, D0 | 16.4 [13.9 to 19.2] | 20.4 [12.5 to 33.2] | 13.7 [9.3 to 20.1]
  H1N1, D21 | 173.5 [146.8 to 205.0] | 211.9 [132.4 to 339.0] | 126.0 [77.0 to 206.3]
  H1N1, D180 | 51.7 [43.9 to 61.1] | 74.2 [48.0 to 114.7] | 45.3 [28.9 to 71.0]
  H3N1, D0 | 16.7 [14.4 to 19.4] | 14.4 [9.8 to 21.2] | 14.6 [10.2 to 20.8]
  H3N1, D21: number analyzed (Participants) | 256 | 37 | 42
  H3N1, D21 | 121.4 [105.1 to 140.2] | 166.0 [108.9 to 253.2] | 166.7 [119.2 to 233.3]
  H3N1, D180 | 42.1 [37.1 to 47.9] | 46.4 [33.9 to 63.7] | 61.9 [44.0 to 87.1]
  BRI, D0 | 31.1 [26.8 to 36.2] | 36.8 [24.8 to 54.5] | 23.8 [16.7 to 33.9]
  BRI, D21 | 179.0 [158.4 to 202.2] | 137.7 [106.0 to 179.0] | 62.9 [43.6 to 90.8]
  BRI, D180 | 120.1 [106.8 to 134.9] | 114.2 [92.9 to 140.4] | 68.4 [49.4 to 94.6]
  FLO, D0 | 77.3 [66.5 to 89.9] | 92.9 [64.6 to 133.7] | 68.4 [47.4 to 98.7]
  FLO, D21 | 399.2 [355.8 to 447.9] | 194.8 [153.5 to 247.2] | 275.8 [194.1 to 392.0]
  FLO, D180 | 253.1 [226.4 to 282.9] | 167.8 [129.2 to 217.8] | 239.6 [171.6 to 334.1]

16. Secondary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥1:40, or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 4 assessed influenza strains were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N1), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 (FLO) flu strains.
Time Frame: At Day 21 (D21) after vaccination.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 1241 | 204 | 211
Participants
  H1N1, D21: number analyzed (Participants) | 1238 | 204 | 211
  H1N1, D21 | 922 | 136 | 138
  H3N1, D21: number analyzed (Participants) | 1237 | 204 | 211
  H3N1, D21 | 823 | 149 | 149
  BRI, D21: number analyzed (Participants) | 1240 | 203 | 210
  BRI, D21 | 685 | 99 | 62
  FLO, D21 | 680 | 68 | 107

17. Secondary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza by Age Strata
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥1:40, or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 4 assessed influenza strains were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N1), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 (FLO) flu strains. Subjects were assessed according to 2 age categories, 18-60Y and ≥ 61Y.
Time Frame: At Day 21 (D21) after vaccination.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 18-60Y Group | GSK2282512A ≥ 61Y Group | Victoria Strain FluLaval 18-60Y Group | Victoria Strain FluLaval ≥ 61Y Group | Yamagata Strain FluLaval 18-60Y Group | Yamagata Strain FluLaval ≥ 61Y Group
Number analyzed (Participants) | 775 | 466 | 127 | 77 | 135 | 76
Participants
  H1N1, D21: number analyzed (Participants) | 775 | 463 | 127 | 77 | 135 | 75
  H1N1, D21 | 616 | 306 | 96 | 40 | 97 | 41
  H3N1, D21: number analyzed (Participants) | 775 | 462 | 127 | 77 | 135 | 76
  H3N1, D21 | 544 | 279 | 99 | 50 | 104 | 45
  BRI, D21: number analyzed (Participants) | 774 | 466 | 126 | 77 | 135 | 75
  BRI, D21 | 522 | 163 | 76 | 23 | 51 | 11
  FLO, D21 | 500 | 180 | 53 | 15 | 88 | 19

18. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease by Age Strata
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0 (i.e. the geometric mean of the within-subject ratios of the Day 21 reciprocal HI titer to the Day 0 reciprocal HI titer). The 4 assessed influenza strains were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N1), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 (FLO) flu strains. Subjects were assessed according to 2 age categories, 18-60Y and ≥ 61Y.
Time Frame: At Day 21 (D21) post vaccination.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK2282512A 18-60Y Group | GSK2282512A ≥ 61Y Group | Victoria Strain FluLaval 18-60Y Group | Victoria Strain FluLaval ≥ 61Y Group | Yamagata Strain FluLaval 18-60Y Group | Yamagata Strain FluLaval ≥ 61Y Group
Number analyzed (Participants) | 775 | 466 | 127 | 77 | 135 | 76
Titer
  SCF - H1N1, D21: number analyzed (Participants) | 775 | 463 | 127 | 77 | 135 | 75
  SCF - H1N1, D21 | 15.8 [14.1 to 17.7] | 7.7 [6.8 to 8.7] | 12.0 [9.2 to 15.6] | 6.0 [4.3 to 8.5] | 11.0 [8.6 to 14.1] | 6.2 [4.3 to 9.0]
  SCF - H3N1, D21: number analyzed (Participants) | 775 | 462 | 127 | 77 | 135 | 76
  SCF - H3N1, D21 | 9.1 [8.3 to 10.1] | 6.0 [5.4 to 6.8] | 12.2 [9.3 to 15.8] | 8.5 [6.1 to 11.8] | 12.0 [9.2 to 15.6] | 6.2 [4.5 to 8.6]
  SCF - BRI, D21: number analyzed (Participants) | 774 | 466 | 126 | 77 | 135 | 75
  SCF - BRI, D21 | 9.5 [8.5 to 10.5] | 3.3 [2.9 to 3.6] | 6.8 [5.3 to 8.7] | 2.4 [1.9 to 3.0] | 3.4 [2.8 to 4.1] | 1.8 [1.4 to 2.3]
  SCF - FLO, D21 | 7.0 [6.3 to 7.7] | 3.2 [3.0 to 3.6] | 3.2 [2.6 to 3.8] | 1.9 [1.5 to 2.3] | 6.3 [5.0 to 8.0] | 2.3 [1.8 to 2.8]

19. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0 (i.e. the geometric mean of the within-subject ratios of the Day 21 reciprocal HI titer to the Day 0 reciprocal HI titer). The 4 assessed influenza strains were the FLU A/California/7/09 (H1N1), FLU A/Victoria/210/09 (H3N1), FLU B/Brisbane/60/08 (BRI) and FLU B/Florida/4/06 (FLO) flu strains.
Time Frame: At Day 21 (D21) post vaccination.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | GSK2282512A Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 1241 | 204 | 211
Titer
  SCF - H1N1, D21: number analyzed (Participants) | 1238 | 204 | 210
  SCF - H1N1, D21 | 12.1 [11.1 to 13.2] | 9.2 [7.5 to 11.4] | 9.0 [7.3 to 11.1]
  SCF - H3N1, D21: number analyzed (Participants) | 1237 | 204 | 211
  SCF - H3N1, D21 | 7.8 [7.2 to 8.5] | 10.6 [8.6 to 13.0] | 9.5 [7.7 to 11.6]
  SCF - BRI, D21: number analyzed (Participants) | 1240 | 203 | 210
  SCF - BRI, D21 | 6.3 [5.8 to 6.9] | 4.6 [3.8 to 5.5] | 2.7 [2.3 to 3.2]
  SCF - FLO, D21 | 5.2 [4.9 to 5.6] | 2.6 [2.3 to 3.0] | 4.4 [3.6 to 5.2]

20. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling at the injection site. Grade 3 pain = significant pain at rest/pain that prevented normal everyday activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within the 7-day (Days 0-6) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects, on subjects for whom results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 417 | 421 | 422 | 208 | 216
Participants
  Any Pain | 260 | 245 | 245 | 93 | 89
  Grade 3 Pain | 9 | 5 | 8 | 2 | 3
  Any Redness | 8 | 11 | 3 | 6 | 3
  Grade 3 Redness | 0 | 0 | 0 | 0 | 0
  Any Swelling | 10 | 13 | 9 | 3 | 8
  Grade 3 Swelling | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (Gastr. Symptoms), headache, muscle ache, shivering, temperature - oral temperature equal to or above (≥) 38.0 degrees Celsius (°C) - and joint pain at location other than the injection site (Joint Pain). Grade 3 temperature = temperature ≥ 39.0 °C. Grade 3 symptom = symptom that prevented normal everyday activity. Related symptom = symptom assessed by the investigator as causally related to study vaccination. Joint pain data were collected for subjects in Canada and Mexico only.
Time Frame: Within the 7-day (Days 0-6) follow-up period after vaccination
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 417 | 421 | 422 | 208 | 216
Participants
  Any Fatigue | 92 | 86 | 93 | 45 | 37
  Grade 3 Fatigue | 6 | 2 | 2 | 2 | 4
  Related Fatigue | 70 | 72 | 78 | 28 | 32
  Any Headache | 93 | 87 | 91 | 41 | 49
  Grade 3 Headache | 4 | 3 | 4 | 1 | 0
  Related Headache | 66 | 60 | 72 | 28 | 35
  Any Muscle Ache | 113 | 105 | 113 | 52 | 40
  Grade 3 Muscle Ache | 2 | 4 | 4 | 1 | 3
  Related Muscle Ache | 93 | 94 | 98 | 39 | 35
  Any Shivering | 39 | 37 | 35 | 16 | 13
  Grade 3 Shivering | 4 | 2 | 2 | 1 | 2
  Related Shivering | 30 | 30 | 27 | 11 | 8
  Any Temperature | 3 | 8 | 8 | 1 | 3
  Grade 3 Temperature | 0 | 3 | 2 | 0 | 1
  Related Temperature | 1 | 8 | 6 | 0 | 2
  Any Joint Pain: number analyzed (Participants) | 196 | 199 | 201 | 102 | 103
  Any Joint Pain | 27 | 27 | 34 | 17 | 15
  Grade 3 Joint Pain: number analyzed (Participants) | 196 | 199 | 201 | 102 | 103
  Grade 3 Joint Pain | 1 | 3 | 1 | 1 | 3
  Related Joint Pain: number analyzed (Participants) | 196 | 199 | 201 | 102 | 103
  Related Joint Pain | 17 | 20 | 21 | 10 | 11
  Any Gastr. | 43 | 35 | 39 | 21 | 16
  Grade 3 Gastr. | 5 | 1 | 4 | 4 | 1
  Related Gastr. | 34 | 26 | 23 | 11 | 8

22. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = any unsolicited AE regardless of intensity or relationship to vaccination. Grade 3 = unsolicited AE that prevented normal everyday activity Related: unsolicited AE assessed by the investigator as related to the vaccination.
Time Frame: Within the 21-day (Days 0-20) follow-up period after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 423 | 424 | 425 | 213 | 218
Participants
  Subject(s) with Any Unsolicited AE(s) | 77 | 80 | 87 | 48 | 51
  Subject(s) with Grade 3 Unsolicited AE(s) | 5 | 5 | 15 | 6 | 7
  Subject(s) with Related Unsolicited AE(s) | 18 | 26 | 21 | 11 | 13

23. Secondary Outcome: Number of Days With Solicited Local Symptoms After Vaccination.
Description: Solicited local symptoms were pain, redness and swelling at the injection site. Analyses of duration for solicited local symptoms were not performed.
Time Frame: Within the 7-day follow-up period after vaccination (Days 0-6)
Population: as for outcome 20
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Days With Solicited General Symptoms After Vaccination
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (Gastr.), headache, muscle ache, shivering, temperature (defined as oral temperature equal to or above 38.0 degrees Celsius) and joint pain at location other than the injection site (Joint Pain). Joint pain data were collected for subjects in Canada and Mexico only. Analyses of duration for solicited general symptoms were not performed.
Time Frame: Within the 7-day follow-up period after vaccination (Days 0-6)
Population: as for outcome 20
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Days With Unsolicited Adverse Events (AEs) After Vaccination
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any: any unsolicited AE regardless of intensity or relationship to vaccination. Grade 3 = unsolicited AE that prevented normal everyday activity. Analyses of duration for unsolicited AEs were not performed.
Time Frame: Within the 21-day (Days 0-20) follow-up period post vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Groups:
- Victoria Strain FluLaval: Subjects received at Day 0 one dose of FluLaval®-VB vaccine containing the Victoria B flu strain. The FluLaval®-VB vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval | Yamagata Strain FluLaval Group
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Reports of solicited local and general adverse events were collected during the 7-day (Days 0-6) follow-up period following vaccination. Reports for serious adverse events were collected throughout the study, from Day 0 to Day 180.
Description: Other Adverse Events were collected only from participants who completed their symptoms sheet.
Groups:
- GSK2282512A 1 Group: Subjects received at Day 0 one dose of the GSK2282512A vaccine, Lot 1. The GSK2282512A vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.dominant arm.
Arm/Group | GSK2282512A 1 Group | GSK2282512A 2 Group | GSK2282512A 3 Group | Victoria Strain FluLaval Group | Yamagata Strain FluLaval Group
Serious Adverse Events (participants affected / at risk) | 15/423 | 13/424 | 7/425 | 3/213 | 7/218
Other Adverse Events (participants affected / at risk) | 294/417 | 286/421 | 284/422 | 127/208 | 113/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2282512A 1 Group (N=423) | GSK2282512A 2 Group (N=424) | GSK2282512A 3 Group (N=425) | Victoria Strain FluLaval Group (N=213) | Yamagata Strain FluLaval Group (N=218)
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Nodal rhythm (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2282512A 1 Group (N=417) | GSK2282512A 2 Group (N=421) | GSK2282512A 3 Group (N=422) | Victoria Strain FluLaval Group (N=208) | Yamagata Strain FluLaval Group (N=216)
Pain (General disorders) | 260 | 245 | 245 | 93 | 89
Fatigue (General disorders) | 92 | 86 | 93 | 45 | 37
Gastrointestinal adverse event(s) (General disorders) | 43 | 35 | 39 | 21 | 15
Headache (General disorders) | 93 | 87 | 91 | 41 | 49
Muscle aches (General disorders) | 113 | 105 | 113 | 52 | 40
Shivering (General disorders) | 39 | 37 | 35 | 16 | 13
Joint pain at other location than injection site (General disorders) | 27 | 27 | 34 | 17 | 15

LIMITATIONS AND CAVEATS:
Analyses of duration for solicited local and general and unsolicited adverse events were not performed. Relationship to vaccination was not computed for medically-attended adverse events. Joint pain data were collected in Canada and Mexico only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.